CLINICAL TRIAL: NCT04063982
Title: Diagnosis-related Outcomes in NeurocriTical Care: Prognostic Estimate by Health-care Providers Versus Risk Scores in Intracerebral and Subarachnoid Hemorrhage
Acronym: DON´T-PERISH
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: German Society of Neurocritical Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: 008/19-ek
Record Dates: First submitted 2019-04-30; First posted 2019-08-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03

CONDITIONS: Intracerebral Hemorrhage; Subarachnoid Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none, only assessment at different time points — assessment at different time points

SUMMARY:
The aim of the observational multicenter trial encompasses the comparison of estimation of the long-term prognosis (functional and cognitive outcomes, quality of life) after intracerebral and subarachnoid hemorrhages assessed by clinical scores, treating physicians and nurses. The scores and the assessment of the treating physicians and nurses are recorded on admission, at 7 and 14 days after symptom onset.

DETAILED DESCRIPTION:
The physicians and nurses responsible for the individual patient's care will be given a questionaire. They are asked to estimate the functional and cognitive status as well as quality of life of their patient. The patient with intracerebral hemorrhage and subarachnoid hemorrhage is examined and assessed with respective established and validated prognostic scores and models at the same time points.

The actual prognosis is assessed by telephone interview and questionaires at 3 and 6 months, either from the patient or his/her caretaker.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracerebral hemorrhage or nontraumatic subarachnoid hemorrhage
* Treatment in Centers with neurocritical care expertise

Exclusion Criteria:

* Language other than German and English
* Restriction of diagnostic and therapeutic measures during acute hospitalization according to advanced directives
* Admission > 48 hours after symptom onset
* Hemorrhage due to trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted with acute spontaneous intracerebral and nontraumatic subarachnoid hemorrhage to a center with neurocritical care expertise
Sampling Method: Non-Probability Sample
Enrollment: 1085 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale dichotomized 0-2 versus 3-6 at 6 months | 6 months
  Modified Rankin Scale dichotomized 0-2 (good functional outcome) versus 3-6 (poor functional outcome)

SECONDARY OUTCOMES:
Modified Rankin Scale dichotomized 0-2 versus 3-6 at 3 months | 3 months
  Modified Rankin Scale dichotomized 0-2 (good functional outcome) versus 3-6 (poor functional outcome)
Modified Rankin Scale dichotomized 0-3 versus 4-6 at 6 months | 6 months
  Modified Rankin Scale dichotomized 0-3 (good functional outcome) versus 4-6 (poor functional outcome)
Modified Rankin Scale dichotomized 0-3 versus 4-6 at 3 months | 3 months
  Modified Rankin Scale dichotomized 0-3 (good functional outcome) versus 4-6 (poor functional outcome)
Quality of life measured by Short Form Health Survey Short Form (SF)-36 | 3 and 6 months
  Short Form Health Survey Short Form (SF)-36: Out of the 36 items, the following 8 subscales/dimensions are assessed and compared to the values of the normal Population: physical function (10 items), physical role function (4 items), physical pain (2 items), general perception of health status (5 items), vitality (4 items), social function and Integration (2 items), emotional role functioning (3 items), psychological well-being (5 items), Change of health status, compared to one year ago (1 item). The first 4 dimensions can be summarized to the physical sum scale, the second 4 items comprise the psychological sum scale.
Quality of life measured by Sickness Impact Profile | 3 and 6 months
  Sickness Impact Profile: 189 items in 14 topic categories. The physical dimension score is obtained by adding the scale values for each item checked within categories body care and movement, mobility, and ambulation, dividing by the maximum possible dysfunction score for these categories, and then multiplying by 100; the psychosocial dimension score is obtained by adding the scale values for each item checked within categories emotional behavior, social interaction, alterness behavior, and communication, dividing by the maximum possible dysfunction score for these categories, and then multiplying by 100. The scores for the remaining categories are always calculated individually. The overall score for the SIP is calculated by adding the scale values for each item checked across all categories and dividing by the maximum possible dysfunction score for the SIP. This figure is then multiplied by 100 to obtain the SIP overall score.
Cognitive outcome Telephone Interview for Cognitive Status | 3 and 6 months
  Telephone Interview for Cognitive Status: During the telephone interview scores for 22 questions are obtained and added to a total score. The qualitative interpretive ranges are 33-41: cognitive impairment unlikely; 26-32 cognitive impairment may be or may not be present dependent on patients's age, education, history, etc.; 21-25: mild cognitive impairment; </=20: moderate to severe cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Katja E Wartenberg, MD, Principal Investigator — University of Leipzig
Locations (10):
- Germany (10):
  - Charité University Hospital, Berlin
  - University Hospital of Duesseldorf, Düsseldorf
  - University of Frankfurt, Frankfurt
  - Wolf-Dirk Niesen, Freiburg im Breisgau
  - University of Leipzig, Leipzig
  - University of Mainz, Mainz
  - Minden Hospital, Minden
  - LMU University of Munich, Munich
  - Osnabrueck Hospital, Osnabrück
  - University Hospital of Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No